CLINICAL TRIAL: NCT03074110
Title: Isocapnic Hyperventilation for Enhancing Recovery After Inhalation Anaesthesia - an Alternative Method
Brief Title: Isocapnic Hyperventilation - an Alternative Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Katarina Hallén, Consultant, Sahlgrenska University Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: GLS-588681
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Oropharyngeal Neoplasms
Keywords: Inhalation Anaesthetics, Sevoflurane; Carbon Dioxide; Hyperventilation; Anaesthesia Recovery Period; Ventilators
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hyperventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isocapnic hyperventilation (Active Comparator): After end of surgery, hyperventilation and administration of a small, precalculated amount of CO2 into the breathing circuit will be performed.
  Interventions: Device: Isocapnic hyperventilation
- Standard procedure (No Intervention): After end of surgery, patients will be subdued to a standard weaning procedure.

INTERVENTIONS:
Device: Isocapnic hyperventilation — Mechanical hyperventilation to enhance elimination of inahalation anesthetics. Administration of a precalculated flow of CO2 according to gender and weight into the inspiratory limb of the breathing circuit in order to avoid hypocapnia.
  Other Names: Normocapnic hyperventilation
  Arms: Isocapnic hyperventilation

SUMMARY:
Isocapnic hyperventilation (IHV) is a method that shortens time to extubation after inhalation anaesthesia by increasing airway carbon dioxide (CO2) during hyperventilation (HV). In two experimental studies (mechanical lung model and porcine model) and in a pilot study on patients undergoing sevoflurane anaesthesia for major ear-nose-throat (ENT) surgery, the investigators evaluated the feasibility of an alternative technique of IHV. By performing a prospective, randomised controlled study, the investigators want to further test this alternative method for IHV.

DETAILED DESCRIPTION:
Isocapnic hyperventilation (IHV) provides an alternative method for weaning from inhalation anaesthesia which decreases the time to eye-opening, extubation and time spent in the PACU. The method is well known since at least 40-50 years and involves the maintenance of a stable CO2 level during hyperventilation, which increases the elimination of anaesthetic gas without producing hypocapnia. Studies have declared that the reduction in time to eye-opening is 50-60 % compared to a standard weaning procedure after inhalation anaesthesia.

There are several principally different ways to maintain the CO2 level during hyperventilation, where a number of technical solutions that add dead-space to the anaesthesia circuit and thereby produce rebreathing of CO2 during hyperventilation are the most studied methods so far. However, the original method of directly adding CO2 to the breathing circuit during hyperventilation could be considered in need of a re-evaluation, as modern anaesthesia delivery units and monitoring equipment to a great extent can eliminate the risk of hypercapnia, that was described with this procedure in the 1980ies.

An alternative IHV method is to directly infuse CO2 to the inspiratory limb of the breathing circuit through a mixing box while using mechanical hyperventilation by a standardised protocol. This technique was recently evaluated by the investigators, in a bench test, and in an in vivo model. Based on these studies, the CO2 dosage needed to achieve isocapnia during HV at various levels of alveolar ventilation, CO2 production and dead space was estimated and a gender- and weight-based nomogram for CO2 delivery during IHV was constructed. Furthermore, the investigators could show, in vivo, that the washout time of sevoflurane anaesthesia was one-third compared to normal ventilation. The feasibility of this IHV method was evaluated in a pilot study in humans, based on the results of our two previous experimental studies. To finalize the project the investigators now conduct a prospective randomized trial to evaluate the efficacy of the method, compared to a standard weaning procedure, after long-term sevoflurane anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for major elective ear-nose-throat (ENT) surgery after informed consent was obtained during the pre-operative evaluation.

Exclusion Criteria:

* Patients with severe pulmonary or circulatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Time to extubation | 5-20 minutes
Time to eye-opening | 10-25 minutes
Time to discharge from OR | 15-40 minutes

SECONDARY OUTCOMES:
Postoperative recovery | 60 minutes
  Postoperative quality of recovery (PQRS) scale
Time to eligible for discharge from post-anaesthesia care unit (PACU) | 1-6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hallen K, Stenqvist O, Ricksten SE, Lindgren S. Isocapnic hyperventilation shortens washout time for sevoflurane - an experimental in vivo study. Acta Anaesthesiol Scand. 2016 Oct;60(9):1261-9. doi: 10.1111/aas.12761. Epub 2016 Jul 10. PMID 27396945
- [Background] Hallen K, Stenqvist O, Ricksten SE, Lindgren S. A simple method for isocapnic hyperventilation evaluated in a lung model. Acta Anaesthesiol Scand. 2016 May;60(5):597-606. doi: 10.1111/aas.12674. Epub 2015 Dec 21. PMID 26688296